CLINICAL TRIAL: NCT06238596
Title: Rehabilitation Intervention to Prevent Adverse Events Related to Androgen-deprivation Therapy (ADT) in Patients With Metastatic Prostate Cancer (PCa): a Single Arm Feasibility Study (ReCaP Study)
Acronym: ReCaP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ReCaP
Record Dates: First submitted 2024-01-25; First posted 2024-02-02 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-06

CONDITIONS: Metastatic Prostate Cancer (PCa) in ADT; Rehabilitation
Keywords: Rehabilitation; feasibility; adverse events
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Rehabilitation

STUDY DESIGN:
Intervention Model Description: This is a drug-free, single arm, single center, superiority, interventional study aimed at treatment feasibility.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- rehabilitation + standard of care (SOC) (Experimental): All enrolled patients will start a supervised rehabilitation program for 12 weeks
  Interventions: Procedure: rehabilitation

INTERVENTIONS:
Procedure: rehabilitation — The rehabilitation intervention will be led by a Physiotherapist and will include: a 12 weeks standardized multicomponent exercise (aerobic, resistance, balance and flexibility, and impact exercise if indicated), supervised by the physiotherapist, on an outpatient basis or in telerehabilitation. This program will be adapted to single patient needs. Every exercise session will last almost 60 minutes and patients will be supervised twice a week. One more exercise session per week will be self-managed by patients.

SUMMARY:
This is a drug-free, single arm, single center, superiority, interventional study aimed at treatment feasibility.

The main aim of the current study is to assess feasibility of a tailored exercise program as measured by adherence to exercise program in metastatic PCa patients undergoing ADT.

Secondary aims are: to deepen the knowledge on other feasibility aspects (recruitment/retention), to monitor safety, to assess the effects in reducing the AEs of ADT (on loss of strength, loss of physical performance and fatigue, number of accidental falls and fractures), to monitor pain and the change in physical activity habits.

The rehabilitation intervention will be led by a Physiotherapist and will include: a 12 weeks standardized multicomponent exercise (aerobic, resistance, balance and flexibility, and impact exercise if indicated), supervised by the physiotherapist, on an outpatient basis or in telerehabilitation. This program will be adapted to single patient needs. Every exercise session will last almost 60 minutes and patients will be supervised twice a week. One more exercise session per week will be self-managed by patients.

At baseline a physiatrist will visit patients with bone metastasis and collect data on sites of bone metastasis, associated level of pain, and risk of pathological fractures. For all participants, the physiotherapist will assess muscle strength (Hand Grip Strength-HGS), physical performance (Short Physical Performance Battery-SPPB), level of fatigue (FACIT-F), and data collection on physical activity habits (International Physical Activity Questionnaire-IPAQ).

The enrollment will be closed after 1 year from the activation of the study or when the target of patients will be reached, whichever occurs firstly.

For each patient, data will be collected for 12 months. The duration of the study is expected to be around 2 years.

Follow-ups are scheduled at 12 weeks, 24 weeks and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of prostatic adenocarcinoma;
* Metastatic disease candidate to ADT treatment and ADT free;
* ECOG PS 0-1.

Exclusion Criteria:

* Physical conditions that may limit adherence to the study (heart failure NYHA 3-4, pathologic fractures, previous disability limiting exercise, etc);
* Psychological/psychiatric conditions that may limit adherence to the study (moderate-severe cognitive impairment, psychiatric disorders, etc.)
* Other concomitant active malignancies

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-09-06 (Actual); Primary Completion 2025-03-03 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
adherence | 12 weeks
  Defined as percentage of patients who complete treatment schedule ≥ 75%

SECONDARY OUTCOMES:
recruitment rate | 12 weeks, 24 weeks, 12 months
  percentage of patients who agree to adhere to the study
retention rates | 12 weeks, 24 weeks, 12 months
  percentage of enrolled patients undergoing re-evaluation at these times
Safety and Tolerability | baseline, 12 weeks, 24 weeks, 12 months
  monitoring of accidental falls, traumatic and pathologic fractures occurred during the study course, and pain in the sites of bone metastasis (measured with NRS Scale); we will distinguish between AEs related to exercise program (pain or falls or fractures occurred during exercise sessions) from AEs not related to exercise;
hand grip strength (HGS) | baseline, 12 weeks, 24 weeks, 12 months
  dichotomized as <27 (low) and >=27Kg (normal)
physical activity (PA) | baseline, 12 weeks, 24 weeks, 12 months
  measured by International Physical Activity Questionnaire (IPAQ)
physical performance | baseline, 12 weeks, 24 weeks, 12 months
  measured by Short Physical Performance Battery (SPPB)
fatigue | 12 weeks, 24 weeks, 12 months
  measured by Functional Assessment of Chronic Illness Therapy - Fatigue Scale (FACIT-F)

CONTACTS AND LOCATIONS:
Locations (1):
- SOC Oncologia Medica Provinciale, Reggio Emilia, Italy, Italy

IPD SHARING:
Plan to Share IPD: No